CLINICAL TRIAL: NCT00542776
Title: Impact of Immunosuppression in Patients With Inflammatory Bowel Disease on Responsiveness to Influenza Vaccine
Brief Title: Impact of Immunosuppression in IBD Patients on Response to Influenza Vaccine
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Ying Lu, MD, Children's Hospital Boston
Other Study IDs: 07-09-0345
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2007-12

CONDITIONS: Inflammatory Bowel Disease (IBD); Immunosuppressed or Non-Immunosuppressed; Influenza Vaccine; Antibody Titers; Seroprotective Titers
Keywords: inflammatory bowel disease (IBD); immunosuppressed or non-immunosuppressed; influenza vaccine; antibody titers; seroprotective titers; vaccine-associated adverse events
MeSH Terms: conditions — Inflammatory Bowel Diseases; Influenza, Human | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for seroprotection rate and antibody titers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: IBD patients on immunosuppressive therapy
  Interventions: Other: blood draw
- 2: IBD patients on non-immunosuppressive therapy (e.g., aminosalicylates, antibiotics) or on no medications
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — drawing blood for seroprotection and antibody titers to the 3 strains of influenza on Day 1 and Month 1 (3-8 weeks)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of influenza vaccine in patients with inflammatory bowel disease (IBD) on immunosuppressive therapy with IBD patients on aminosalicylates and healthy historical controls.

DETAILED DESCRIPTION:
Influenza is an extremely contagious airborne disease caused by influenza viruses. It can cause mild to severe illness, and even death. Patients who have inflammatory bowel disease (IBD) have a higher risk of getting serious complications if they are infected. Current guidelines recommend the influenza vaccine for IBD patients. However, many IBD patients take immunosuppressive agents and we are uncertain as to their capacity to mount a truly protective response after vaccination. This is an important area of research because if IBD patients do not have an adequate immunological response, then we may need to enhance their response by increasing the dosage or giving booster shots.

Many clinicians who treat patients with autoimmune diseases are asking if the vaccine is safe and effective. Many IBD patients will receive the vaccine without proper studies being performed to answer these questions. The study we are proposing has important clinical and public health significance. It is a step toward answering the question whether vaccination with the influenza vaccine is safe in patients with IBD and if patients on different types of immunosuppressive medications respond similarly and if they respond as well as healthy controls to the vaccine. There are more than one million people in the United States who have been diagnosed with IBD. Thus, the information gained from this clinical study will provide important knowledge to physicians caring for immunocompromised patients who are considering vaccination.

Studies on the immunological response of immunocompromised patients (e.g., transplant, HIV, oncology, chronic renal failure, SLE) to the influenza vaccine have demonstrated that some of these patients develop antibody titers at a protective level within 4-6 weeks. However, the titers were decreased compared to healthy controls, especially if the immunocompromised patients were on immunosuppressive agents. The frequency of influenza in immunocompromised patients was lower after immunization and there were almost no major side effects from the vaccine.

There is little data on immune response to vaccination in children with IBD. One recently published study compared influenza titers before and after vaccination among 3 pediatric groups: IBD patients who received immunosuppressive therapy, IBD patients who did not receive immunosuppressive therapy, and healthy controls. All IBD patients in the study had a decrease in response to one of three influenza strains when compared to controls. IBD patients who received both immunomodulators and infliximab had a lower immune response rate to two influenza strains when compared to controls. There was no difference in immune response among IBD patients on immunomodulators only, IBD patients on ASA, and controls. There was no difference in rates of adverse events between IBD patients and controls

The primary aim of this research are to measure seroprotection in IBD patients who are on or off immunosuppressive agents after receiving the influenza vaccine. The hypothesis is that IBD patients on immunosuppression have impaired immunity, and therefore, will have a lower seroprotection rate after immunization compared to IBD patients not on immunosuppression. If data is available, we will also compare each group to historical healthy controls given the same vaccine. The secondary aims are to determine the antibody titer levels and side effects these patients have.

The patient population includes IBD patients who are off immunosuppression and IBD patients who are on immunosuppression. Recruiting approximately 75 patients per group will provide adequate power for the study. A blood sample will be taken from all IBD patients to evaluate baseline antibody levels and markers (e.g., CBC, ESR, albumin) before or immediately after immunization with the influenza vaccine. Lab tests will be redrawn at Month 1 (3-8 weeks) to evaluate the level of antibody titers and follow the markers. During the study, we will track basic laboratory measures, disease status by using the Pediatric Crohn's Disease Active Index or Modified Harvey-Bradshaw Score for UC, side effects and adverse events from the vaccinations.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease, ulcerative colitis, or indeterminate colitis diagnosed by standard clinical, radiographic, endoscopic, and histologic criteria.
2. Age 5 years and older
3. Actively or previously followed by a gastroenterologist at Children's Hospital Boston
4. On non-immunosuppressants (aminosalicylates, antibiotics, or no medications) and/or immunosuppressants (steroids, immunomodulators, TNF-alpha inhibitors) for the past 30 days. Standard concomitant medications (e.g. antihistamines, acetaminophen) will be allowed.

Exclusion Criteria:

1. History of bleeding disorder that would make hematoma likely (eg hemophilia, von Willebrand's disease)
2. Received influenza vaccination during the current influenza season
3. Contraindications to the influenza vaccine (such as severe allergic reaction to prior influenza vaccine)
4. Fever within 48 hr prior to injection
5. Receipt of another vaccination within 2 days of influenza vaccine dose (and no other vaccines planned for 2 days after influenza vaccine)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 5 years and older with documented inflammatory bowel disease (Crohn's disease, ulcerative colitis, indeterminate colitis)
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
seroprotection rate | 3-8 weeks after vaccination

SECONDARY OUTCOMES:
vaccine-associated adverse events | up to 8 weeks after vaccination
antibody titer levels | 3-8 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Blumberg EA, Albano C, Pruett T, Isaacs R, Fitzpatrick J, Bergin J, Crump C, Hayden FG. The immunogenicity of influenza virus vaccine in solid organ transplant recipients. Clin Infect Dis. 1996 Feb;22(2):295-302. doi: 10.1093/clinids/22.2.295. PMID 8838186
- [Background] Soesman NM, Rimmelzwaan GF, Nieuwkoop NJ, Beyer WE, Tilanus HW, Kemmeren MH, Metselaar HJ, de Man RA, Osterhaus AD. Efficacy of influenza vaccination in adult liver transplant recipients. J Med Virol. 2000 May;61(1):85-93. PMID 10745238
- [Background] Banic S, Koren S, Tomazic J, Vidmar L, Ihan A, Poljak M, Avsic-Zupanc A. Influenza vaccination of human immunodeficiency virus 1-infected patients receiving antiretroviral therapy. Acta Virol. 2001 Feb;45(1):39-44. PMID 11394576
- [Background] Matsuzaki A, Suminoe A, Koga Y, Kinukawa N, Kusuhara K, Hara T. Immune response after influenza vaccination in children with cancer. Pediatr Blood Cancer. 2005 Nov;45(6):831-7. doi: 10.1002/pbc.20470. PMID 16007602
- [Background] Cavdar C, Sayan M, Sifil A, Artuk C, Yilmaz N, Bahar H, Camsari T. The comparison of antibody response to influenza vaccination in continuous ambulatory peritoneal dialysis, hemodialysis and renal transplantation patients. Scand J Urol Nephrol. 2003;37(1):71-6. doi: 10.1080/00365590310008749. PMID 12745749
- [Background] Suga T, Niki H, Niikura M, Matsumoto Y, Nishimura T, Nakajima K, Miyazaki M, Endoh M, Nomoto Y, Sakai H. Influenza antibody titers after vaccination of chronic renal failure patients; before and during hemodialysis, or on continuous ambulatory peritoneal dialysis. Tokai J Exp Clin Med. 1990 May;15(2-3):245-51. PMID 2130531
- [Background] Holvast A, Huckriede A, Wilschut J, Horst G, De Vries JJ, Benne CA, Kallenberg CG, Bijl M. Safety and efficacy of influenza vaccination in systemic lupus erythematosus patients with quiescent disease. Ann Rheum Dis. 2006 Jul;65(7):913-8. doi: 10.1136/ard.2005.043943. Epub 2005 Dec 1. PMID 16322083
- [Background] Abu-Shakra M, Press J, Varsano N, Levy V, Mendelson E, Sukenik S, Buskila D. Specific antibody response after influenza immunization in systemic lupus erythematosus. J Rheumatol. 2002 Dec;29(12):2555-7. PMID 12465151
- [Background] Mamula P, Markowitz JE, Piccoli DA, Klimov A, Cohen L, Baldassano RN. Immune response to influenza vaccine in pediatric patients with inflammatory bowel disease. Clin Gastroenterol Hepatol. 2007 Jul;5(7):851-6. doi: 10.1016/j.cgh.2007.02.035. Epub 2007 Jun 4. PMID 17544875